CLINICAL TRIAL: NCT04245657
Title: Investigation of the Factors of Hang-Grip Strength-related Upper Extremity Functionality After Breast Cancer Surgery
Brief Title: Factors Affecting Functionality in Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Alper Tuğral, Alper Tuğral, PT, MSc, Lecturer. Izmir Bakircay University Faculty of Health Sciences, Department of Physical Therapy and Rehabilitation, Izmir Bakircay University
Other Study IDs: BakircayU
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer; Breast Cancer Female; Breast Cancer Lymphedema; Breast Carcinoma in Situ; Hand Grasp; Pain, Shoulder
Keywords: Breast Cancer; Lymphedema; Upper Extremity Function; Hand Grip Strength
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema; Breast Carcinoma In Situ; Shoulder Pain; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Survivors: Female breast cancer survivors who underwent unilateral breast cancer surgery ( total or conservative) and completed their adjuvant therapies such as chemotherapy and radiotherapy prior to participation in this study.
  Interventions: Other: Tissue Dielectric Constant Measurement; Other: Muscle strength measurement; Other: Hand-Grip Strength Measurement; Other: Pain Threshold Measurement; Other: International Physical Activity Questionnaire-Short Form (IPAQ-SF); Other: Fatigue Impact Scale; Other: Disabilities of Arm, Shoulder and Hand Scale (DASH); Other: Exercise Benefits/ Barriers Scale; Other: Beck Depression Scale

INTERVENTIONS:
Other: Tissue Dielectric Constant Measurement — Sub-tissue fluid proportion will be evaluated via Moisture Meter D (Delfin Technologies, Kuopio, Finland) on both upper extremity (right and left) in predefined reference points on volar side (6 cm distal and 8 cm proximal points from cubital crease, 10 cm inferior side point from axilla and dorsal point of web space in the hand) by using four different probes which can assess 0.5 mm, 1.5 mm, 2.5 mm and 5.0 mm depth. Values taken by 2.5 mm depth probe will be used to calculate the ratio (affected side TDC value/Unaffected side TDC value) to stage lymphedema severity along with the International Society of Lymphology staging system. This device mainly aims to assess the dielectric constant of tissues which is related to the amount of tissue water. In the case of pre-lymphedema or lymphedema, one can assess objectively regarding sub-tissue fluid changes via this device. Triplicate measurements will be taken for each reference point.
Other: Muscle strength measurement — Participants' muscle strength of shoulder flexion, abduction, and elbow flexion will be assessed via Handheld digital dynamometer (Lafayette Manual Muscle Tester, Model 01165, LaFayette Instruments, NY, USA). Both upper extremities will be assessed three times and the average value will be recorded.
Other: Hand-Grip Strength Measurement — Handgrip strength will be assessed with LaFayette Professional Hand Dynamometer, Model 5030L1, LaFayette Instruments, NY, USA). The standard position which can be achieved by 90-degree elbow flexion, shoulder abducted, and hand mid-prone positioned; 90-degree shoulder abduction and 90-degree shoulder abduction positions will be used to assess hang-grip strength. Three measurements will be requested and the maximum value of them will be recorded. 1 minute resting period will be provided between the positions at which handgrip is assessed.
Other: Pain Threshold Measurement — The sensitive pain threshold and normal pain threshold will be evaluated by a digital algometer (Wagner FDIX, Greenwich, USA) on reference points as follows: C5-C6 zygapophyseal joints' lateral points, upper trapezius (proximal, middle and distal lateral points, length measured by a tape from C7 Processus spinosus to acromion and this length will be divided equally into three parts for proximal, middle and distal lateral point), deltoid muscle (crista deltoidea), dorsum of the webspace.
Other: International Physical Activity Questionnaire-Short Form (IPAQ-SF) — This scale was intended to be filled to assess participants' physical activity levels within the last seven days. Then, MET calculations will be done via a basic Excel Spreadsheet which is pre-defined MET values formulated inside. Scale data then obtained according to the participants' answers and recorded.
Other: Fatigue Impact Scale — This scale has 9 items that can be answered as "Strongly Disagree" through "Strongly Agree" by numbered as 1 and 7, respectively. Then total points will be calculated and divided into 9 to achieve the Fatigue Impact Scale score. The higher points will be indicated more perceived fatigue, while lower points indicate less.
Other: Disabilities of Arm, Shoulder and Hand Scale (DASH) — DASH has 30 items related to upper extremity function. Participants will be requested to grade some expressions related to the function within a 5-point Likert scale as follows: "No difficulty: 1, Mild Difficulty:2, Moderate Difficulty: 3, Severe Difficulty: 4 and Unable to perform: 5). The symptom score of the DASH will be calculated as dividing filled items total score to filled items' number and minus one from this data then multiplying with 25. The higher points indicate a deteriorated shoulder and hand function while lower points indicate a better upper extremity function.
Other: Exercise Benefits/ Barriers Scale — Exercise Benefits/Barriers Scale has 43 items each can be graded within a four-point Likert type scale. Barrier items are reverse coded. 43 items are all related to exercise and exercise beliefs in both in the aspect of health and general. Strongly disagree, disagree, agree, strongly agree will be scored as 1,2,3,4 or vice versa whether the item should de reversely coded, respectively. Total scores ranged between 29 and 172. The barrier scale score is ranged between 14 and 56. The benefits scale is also ranged between 29 and 116. The higher the score of Barriers scale, the greater the perception of barriers to exercise.
Other: Beck Depression Scale — Beck Depression Scale has 21 items each can be scored within 0 to 3. All items are related to the depressive mood of a participant. The higher the score of the Beck Depression Scale, the higher the depression level.

SUMMARY:
Breast cancer is the most frequent cancer type in women globally. In conjunction with the new developments, breast cancer survival has increased therefore the management of long-term complications has gained importance. Breast cancer survivors can face the loss of muscle strength, increased fatigue and diminished physical function associated with treatment-related long term effects and psychological affection and thereby reduced quality of life. Upper extremity lymphedema or breast cancer-related lymphedema (BCRL) is one of the most prominent long term complications which affects breast cancer survivors in many ways after breast cancer surgery. It has been reported that breast cancer survivors with BCRL have the lower muscle strength and more activity limitations when compared to the ones free of BCRL. In BCRL, affected extremity has been found to 36% more weaker when compared to the unaffected side. Fatigue is one of the most prominent symptoms when considering cancer-related symptoms in cancer survivors. It has been stated that increased fatigue is correlated with increased activity limitation and deterioration in physical function. The hand-grip test which is frequently used in the assessment of decreased muscle function has been stated as a reliable and repeatable test in breast cancer survivors. In addition, this test is frequently applicable to assess mortality, physical and functional capacity, symptoms after surgery and to designate an exercise program. There are studies that investigate upper extremity function associated with hang-grip strength in breast cancer survivors. Yet, there is a lack of the objective result or conclusion of the BCRL effect on upper extremity function which is assessed with hang-grip strength when compared without BCRL. Therefore, this study is planned to investigate of cumulative effects of factors such as lymphedema severity, age, fatigue, body mass index, muscle strength, physical activity level, pain level, exercise benefits/barriers scale score on hand-grip strength related upper extremity functionality in breast cancer survivors.

DETAILED DESCRIPTION:
Investigation of the Factors of Hand-Grip Strength-related Upper Extremity Functionality in Breast Cancer Survivors

Breast cancer is the most frequent cancer type in women globally. In the United States, there are almost 3 million breast cancer cases and this number gradually increasing in recent years. In conjunction with the new developments, breast cancer survival has increased therefore the management of long-term complications has gained importance. Breast cancer survivors can face the loss of muscle strength, increased fatigue and diminished physical function associated with treatment-related long term effects and psychological affection and thereby reduced quality of life. In addition to the reduced quality of life, breast cancer survivors experience reduced and altered upper extremity function. The Data not only reported by breast cancer survivors but also derived by objective assessment tools state that the high prevalence of disrupted upper extremity function. Studies reported that the deterioration of shoulder function and reduced strength and flexibility in the range of between 16% to 43%, however, these parameters followed a stabile pattern within a year while some parameters which are assessed relatively in short periods were found in higher prevalence. In addition to these, reduced mobility of head and neck, perceived fatigue, reduced upper extremity strength are factors that induce functional limitations in breast cancer survivors.

Upper extremity lymphedema or breast cancer-related lymphedema (BCRL) is one of the most prominent long term complications which affects breast cancer survivors in many ways after breast cancer surgery. Lymphedema is characterized by the inability of the function of the lymphatic system which can result in the accumulation of protein-rich lymphatic fluid in interstitial spaces in addition to skin changes in related body regions and extremities. Untreated lymphedema causes chronic inflammation, cellulitis, pain, fatigue, cosmetic deformity, restriction in mobility and related problems and therefore ineffective usage of the extremity concerning diminished functionality has occurred. It is known that the esthetical concern and emotional stress manifested by lymphedema cause deterioration in physical function. The heaviness feeling, fibrosis and skin infections caused by lymphedema not only can increase psychological stress but also induce musculoskeletal complications in the long term. It has been reported that breast cancer survivors with BCRL have the lower muscle strength and more activity limitations when compared to the ones free of BCRL. In BCRL, affected extremity has been found to 36% more weaker when compared to the unaffected side. Through augmented severity and stage of lymphedema, reduced physical functions are taken place in the clinical condition. Patients without BCRL can increase their cumulative musculoskeletal problems by avoiding physical activity and exercise due to misguidance and fear of lymphedema while the ones with BCRL have to fear the increased severity of lymphedema by doing so. Lymphedema can bring with problems such as reduced physical activity and weight gain thereby constitution of the basis of functional limitations is settled.

Increased fat mass and body mass index are reported in the range of 50% to %96 in breast cancer survivors. Optimal upper extremity function is important for maintaining an independent daily life and day routines and to perform works that need physical strength in terms of the general quality of life. However, affecting factors and incidence of their impact on upper extremity function in the aspect of physical, functional and psychological are still have been the research issue. The literature reports that the frequently reduced muscle strength due to cancer-related symptoms along with the altered motor control in shoulder and neck musculature. Fatigue is one of the most prominent symptoms when considering cancer-related symptoms in cancer survivors. It has been stated that increased fatigue is correlated with increased activity limitation and deterioration in physical function. The hand-grip test which is frequently used in the assessment of decreased muscle function has been stated as a reliable and repeatable test in breast cancer survivors. Besides, this test is frequently applicable to assess mortality, physical and functional capacity, symptoms after surgery and to designate an exercise program.

Some studies investigate upper extremity function associated with handgrip strength in breast cancer survivors. Yet, there is a lack of the objective result or conclusion of the BCRL effect on upper extremity function which is assessed with hang-grip strength when compared without BCRL. Therefore, this study is planned to investigate of cumulative effects of factors such as lymphedema severity, age, fatigue, body mass index, muscle strength, physical activity level, pain level, exercise benefits/barriers scale score on hand-grip strength related upper extremity functionality in breast cancer survivors.

The primary purpose of this study:

This study is planned to investigate of cumulative effects of factors such as lymphedema severity, age, fatigue, body mass index, muscle strength, physical activity level, pain level, exercise benefits/barriers scale score on hand-grip strength related upper extremity functionality in breast cancer survivors.

Secondary aim:

Which of the aforementioned parameters has the most prominent effect on hand-grip strength related upper extremity functionality in breast cancer survivors

Primary endpoint:

Having reached to a targeted number of breast cancer survivors compatible with the incl/excl criteria of this study

Secondary endpoint:

According to the pilot test result, elimination of parameters that are not significant in the statistical model will be excluded and power analysis will be re-performed. If the current number of the targeted population has been achieved (by achieving at least 80% power, 95% CI), then the study will be finished to save time and resources.

Center: Single-center study

Time range: December 2019- October 2020

Methods:

109 women aged between 25 and 65 years who had unilateral breast cancer surgery will be included in this study (Sample size was determined according to the 0.15 effect size, 80% power, and 95% confidence interval). Within the context of this study, an evaluation form that assesses demographic information (Both patient and clinical demographics such as Name, age, contact information and/or body mass index, time spent after surgery, surgery type, etc) will be requested to fill. Within this form, having lymphedema (yes/no), drug use (especially tamoxifen, yes/no), pain assessment (via visual analog scale), adjuvant therapies (radiotherapy, chemotherapy, yes/no, number of sessions, etc) and shoulder range of motion assessment via goniometer will be evaluated and recorded to the assessment form.

Tissue Dielectric Constant Measurement:

Sub-tissue fluid proportion will be evaluated via Moisture Meter D (Delfin Technologies, Kuopio, Finland) on both upper extremity (right and left) in predefined reference points on volar side (6 cm distal and 8 cm proximal points from cubital crease, 10 cm inferior side point from axilla and dorsal point of web space in the hand) by using four different probes which can assess 0.5 mm, 1.5 mm, 2.5 mm and 5.0 mm depth. Values taken by 2.5 mm depth probe will be used to calculate the ratio (affected side TDC value/Unaffected side TDC value) to stage lymphedema severity along with the International Society of Lymphology staging system.

Muscle strength Participants' muscle strength of shoulder flexion, abduction, and elbow flexion will be assessed via Handheld digital dynamometer (Lafayette Manual Muscle Tester, Model 01165, LaFayette Instruments, NY, USA). Both upper extremities will be assessed three times and the average value will be recorded.

Hand-Grip Strength Handgrip strength will be assessed with LaFayette Professional Hand Dynamometer, Model 5030L1, LaFayette Instruments, NY, USA). The standard position which can be achieved by 90-degree elbow flexion, shoulder abducted, and hand mid-prone positioned; 90-degree shoulder abduction and 90-degree shoulder abduction positions will be used to assess hang-grip strength. Three measurements will be requested and the maximum value of them will be recorded.

Pain Threshold Measurement The sensitive pain threshold and normal pain threshold will be evaluated by a digital algometer (Wagner FDIX, Greenwich, USA) on reference points as follows: C5-C6 zygapophyseal joints' lateral points, upper trapezius (proximal, middle and distal lateral points, length measured by a tape from C7 Processus spinosus to acromion and this length will be divided equally into three parts for proximal, middle and distal lateral point), deltoid muscle (deltoid tuberosity), dorsum of the webspace. Measurements will te took both for right and left upper extremity. Units will be recorded as kgf.

Scales and Forms There will be scales and form which are required to fill out by participants. The following list of scales will be filled with participants themselves.

International Physical Activity Questionnaire-Short Form (IPAQ-SF):

This scale was intended to be filled to assess participants' physical activity levels within the last seven days. Then, MET calculations will be done via a basic Excel Spreadsheet which is pre-defined MET values formulated inside. Scale data then obtained according to the participants' answers and recorded.

Fatigue Impact Scale:

This scale has 9 items that can be answered as "Strongly Disagree" through "Strongly Agree" by numbered as 1 and 7, respectively. Then total points will be calculated and divided into 9 to achieve the Fatigue Impact Scale score. The higher points will be indicated more perceived fatigue, while lower points indicate less.

Disabilities of Arm, Shoulder and Hand Scale (DASH):

DASH has 30 items related to upper extremity function. Participants will be requested to grade some expressions related to the function within a 5-point Likert scale as follows: "No difficulty: 1, Mild Difficulty:2, Moderate Difficulty: 3, Severe Difficulty: 4 and Unable to perform: 5). The symptom score of the DASH will be calculated as dividing filled items total score to filled items' number and minus one from this data then multiplying with 25. The higher points indicate a deteriorated shoulder and hand function while lower points indicate a better upper extremity function.

Exercise Benefits/ Barriers Scale Exercise Benefits/Barriers Scale has 43 items each can be graded within a four-point Likert type scale. Barrier items are reverse coded. 43 items are all related to exercise and exercise beliefs in both in the aspect of health and general. Strongly disagree, disagree, agree, strongly agree will be scored as 1,2,3,4 or vice versa whether the item should de reversely coded, respectively. Total scores ranged between 29 and 172. The barrier scale score is ranged between 14 and 56. The benefits scale is also ranged between 29 and 116. The higher the score of Barriers scale, the greater the perception of barriers to exercise.

Beck Depression Scale

Beck Depression Scale has 21 items each can be scored within 0 to 3. All items are related to the depressive mood of a participant. The higher the score of the Beck Depression Scale, the higher the depression level.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 25 and 65 years old
* Having the ability to read and write in the Turkish language
* Having unilateral (right or left) breast cancer surgery history
* Being a woman
* Finished adjuvant therapies such as chemotherapy and radiotherapy prior to participation

Exclusion Criteria:

* Active infection
* Active/recurrent malignity
* Having orthopedic and/or neurological defect
* Having an advanced postural deficiency
* Having nerve injury (Ulnar, median, radial nerve)
* Having a loss of sensory
* Bilateral (both side) breast cancer surgery
* Having mental and cognitive problems which can interfere to participate
* Serious range of movement restriction in shoulder, elbow and/or wrist joints
* Having Carpal Tunnel Syndrome
* Having reflex denervation and abnormal neural findings

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Being a woman and having the right or left unilateral breast cancer surgery
Study Population: Female Breast cancer survivors aged 25-65 years old who had unilateral breast cancer surgery will be enrolled to this study.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Hand-Grip Strength | 15 minutes
  Handgrip strength will be assessed with LaFayette Professional Hand Dynamometer, Model 5030L1, LaFayette Instruments, NY, USA). The standard position which can be achieved by 90-degree elbow flexion, shoulder abducted, and hand mid-prone positioned; 90-degree shoulder abduction and 90-degree shoulder abduction positions will be used to assess hang-grip strength. Three measurements will be requested and the maximum value of them will be recorded. 1 minute resting period will be provided between the positions at which handgrip is assessed.

SECONDARY OUTCOMES:
Tissue Dielectric Constant Measurement: | 30 minutes
  Sub-tissue fluid proportion will be evaluated via Moisture Meter D (Delfin Technologies, Kuopio, Finland) on both upper extremity (right and left) in predefined reference points on volar side (6 cm distal and 8 cm proximal points from cubital crease, 10 cm inferior side point from axilla and dorsal point of web space in the hand) by using four different probes which can assess 0.5 mm, 1.5 mm, 2.5 mm and 5.0 mm depth. Values taken by 2.5 mm depth probe will be used to calculate the ratio (affected side TDC value/Unaffected side TDC value) to stage lymphedema severity along with the International Society of Lymphology staging system.
Muscle strength | 10 minutes
  Participants' muscle strength of shoulder flexion, abduction, and elbow flexion will be assessed via Handheld digital dynamometer (Lafayette Manual Muscle Tester, Model 01165, LaFayette Instruments, NY, USA). Both upper extremities will be assessed three times and the average value will be recorded. 1 minute resting period will be provided between the positions at which muscle strength is assessed.
Pain Threshold Measurement | 8 minutes
  The sensitive pain threshold and normal pain threshold will be evaluated by a digital algometer (Wagner FDIX, Greenwich, USA) on reference points as follows: C5-C6 zygapophyseal joints' lateral points, upper trapezius (proximal, middle and distal lateral points, length measured by a tape from C7 Processus spinosus to acromion and this length will be divided equally into three parts for proximal, middle and distal lateral point), deltoid muscle (crista deltoidea), dorsum of the webspace. Measurements will te took both for right and left upper extremity. Units will be recorded as kgf.
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | 3 minutes
  This scale was intended to be filled to assess participants' physical activity levels within the last seven days. Then, MET calculations will be done via a basic Excel Spreadsheet which is pre-defined MET values formulated inside. Scale data then obtained according to the participants' answers and recorded.
Fatigue Impact Scale | 3 minutes
  This scale has 9 items that can be answered as "Strongly Disagree" through "Strongly Agree" by numbered as 1 and 7, respectively. Then total points will be calculated and divided into 9 to achieve the Fatigue Impact Scale score. The higher points will be indicated more perceived fatigue, while lower points indicate less.
Disabilities of Arm, Shoulder and Hand Scale (DASH) | 10 minutes
  DASH has 30 items related to upper extremity function. Participants will be requested to grade some expressions related to the function within a 5-point Likert scale as follows: "No difficulty: 1, Mild Difficulty:2, Moderate Difficulty: 3, Severe Difficulty: 4 and Unable to perform: 5). The symptom score of the DASH will be calculated as dividing filled items total score to filled items' number and minus one from this data then multiplying with 25. The higher points indicate a deteriorated shoulder and hand function while lower points indicate a better upper extremity function.
Exercise Benefits/ Barriers Scale | 20 minutes
  Exercise Benefits/Barriers Scale has 43 items each can be graded within a four-point Likert type scale. Barrier items are reverse coded. 43 items are all related to exercise and exercise beliefs in both in the aspect of health and general. Strongly disagree, disagree, agree, strongly agree will be scored as 1,2,3,4 or vice versa whether the item should de reversely coded, respectively. Total scores ranged between 29 and 172. The barrier scale score is ranged between 14 and 56. The benefits scale is also ranged between 29 and 116. The higher the score of Barriers scale, the greater the perception of barriers to exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Yeşim Bakar, Professor, Study Director — Bakırçay University, Fac. of Health Sci, Dept. of Physical Therapy and Rehab; İlker Kızıloğlu, MD, Principal Investigator — İzmir Çiğli State Training Hospital, Department of General Surgery; Alper Tuğral, PT, Principal Investigator — Bakırçay University, Fac. of Health Sci, Dept. of Physical Therapy and Rehab
Locations (1):
- İzmir Çiğli State Training Hospital, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Angelis R, Tavilla A, Verdecchia A, Scoppa S, Hachey M, Feuer EJ, Mariotto AB. Breast cancer survivors in the United States: geographic variability and time trends, 2005-2015. Cancer. 2009 May 1;115(9):1954-66. doi: 10.1002/cncr.24217. PMID 19248047
- [Background] Fong DY, Ho JW, Hui BP, Lee AM, Macfarlane DJ, Leung SS, Cerin E, Chan WY, Leung IP, Lam SH, Taylor AJ, Cheng KK. Physical activity for cancer survivors: meta-analysis of randomised controlled trials. BMJ. 2012 Jan 30;344:e70. doi: 10.1136/bmj.e70. PMID 22294757
- [Background] Satariano WA, Ragland DR, DeLorenze GN. Limitations in upper-body strength associated with breast cancer: a comparison of black and white women. J Clin Epidemiol. 1996 May;49(5):535-44. doi: 10.1016/0895-4356(95)00565-x. PMID 8636727
- [Background] Armer JM. The problem of post-breast cancer lymphedema: impact and measurement issues. Cancer Invest. 2005;23(1):76-83. PMID 15779870
- [Background] Smoot B, Wong J, Cooper B, Wanek L, Topp K, Byl N, Dodd M. Upper extremity impairments in women with or without lymphedema following breast cancer treatment. J Cancer Surviv. 2010 Jun;4(2):167-78. doi: 10.1007/s11764-010-0118-x. Epub 2010 Apr 7. PMID 20373044
- [Background] Lee D, Hwang JH, Chu I, Chang HJ, Shim YH, Kim JH. Analysis of factors related to arm weakness in patients with breast cancer-related lymphedema. Support Care Cancer. 2015 Aug;23(8):2297-304. doi: 10.1007/s00520-014-2584-6. Epub 2015 Jan 10. PMID 25576430
- [Background] Nesvold IL, Reinertsen KV, Fossa SD, Dahl AA. The relation between arm/shoulder problems and quality of life in breast cancer survivors: a cross-sectional and longitudinal study. J Cancer Surviv. 2011 Mar;5(1):62-72. doi: 10.1007/s11764-010-0156-4. Epub 2010 Oct 23. PMID 20972640
- [Background] Garabeli Cavalli Kluthcovsky AC, Urbanetz AA, de Carvalho DS, Pereira Maluf EM, Schlickmann Sylvestre GC, Bonatto Hatschbach SB. Fatigue after treatment in breast cancer survivors: prevalence, determinants and impact on health-related quality of life. Support Care Cancer. 2012 Aug;20(8):1901-9. doi: 10.1007/s00520-011-1293-7. Epub 2011 Oct 13. PMID 21994001
- [Background] Wilmoth MC, Coleman EA, Smith SC, Davis C. Fatigue, weight gain, and altered sexuality in patients with breast cancer: exploration of a symptom cluster. Oncol Nurs Forum. 2004 Nov 16;31(6):1069-75. doi: 10.1188/04.ONF.1069-1075. PMID 15547630
- [Background] Winters-Stone KM, Bennett JA, Nail L, Schwartz A. Strength, physical activity, and age predict fatigue in older breast cancer survivors. Oncol Nurs Forum. 2008 Sep;35(5):815-21. doi: 10.1188/08.ONF.815-821. PMID 18765328
- [Background] Cantarero-Villanueva I, Fernandez-Lao C, Fernandez-DE-Las-Penas C, Diaz-Rodriguez L, Sanchez-Cantalejo E, Arroyo-Morales M. Associations among musculoskeletal impairments, depression, body image and fatigue in breast cancer survivors within the first year after treatment. Eur J Cancer Care (Engl). 2011 Sep;20(5):632-9. doi: 10.1111/j.1365-2354.2011.01245.x. Epub 2011 Mar 17. PMID 21410803
- [Background] Galiano-Castillo N, Fernandez-Lao C, Cantarero-Villanueva I, Fernandez-de-Las-Penas C, Menjon-Beltran S, Arroyo-Morales M. Altered pattern of cervical muscle activation during performance of a functional upper limb task in breast cancer survivors. Am J Phys Med Rehabil. 2011 May;90(5):349-55. doi: 10.1097/PHM.0b013e318214e406. PMID 21765253
- [Background] Vardar-Yagli N, Sener G, Saglam M, Calik-Kutukcu E, Arikan H, Inal-Ince D, Savci S, Altundag K, Kutluk T, Ozisik Y, Kaya EB. Associations among physical activity, comorbidity, functional capacity, peripheral muscle strength and depression in breast cancer survivors. Asian Pac J Cancer Prev. 2015;16(2):585-9. doi: 10.7314/apjcp.2015.16.2.585. PMID 25684491
- [Background] Fernandez-Lao C, Cantarero-Villanueva I, Fernandez-de-las-Penas C, Del-Moral-Avila R, Menjon-Beltran S, Arroyo-Morales M. Widespread mechanical pain hypersensitivity as a sign of central sensitization after breast cancer surgery: comparison between mastectomy and lumpectomy. Pain Med. 2011 Jan;12(1):72-8. doi: 10.1111/j.1526-4637.2010.01027.x. Epub 2010 Dec 10. PMID 21143767
- [Background] Dibai-Filho AV, de Jesus Guirro RR, Koga Ferreira VT, Kelly de Oliveira A, Maria de Almeida A, de Oliveira Guirro EC. Analysis of chronic myofascial pain in the upper trapezius muscle of breast cancer survivors and women with neck pain. J Bodyw Mov Ther. 2018 Apr;22(2):237-241. doi: 10.1016/j.jbmt.2017.04.012. Epub 2017 Apr 28. PMID 29861213
- [Background] Park SW, Lee I, Kim JI, Park H, Lee JD, Uhm KE, Hwang JH, Lee ES, Jung SY, Park YH, Lee JY. Factors associated with physical activity of breast cancer patients participating in exercise intervention. Support Care Cancer. 2019 May;27(5):1747-1754. doi: 10.1007/s00520-018-4427-3. Epub 2018 Aug 25. PMID 30145738
- [Background] Perez CS, das Neves LMS, Vacari AL, de Cassia Registro Fonseca M, de Jesus Guirro RR, de Oliveira Guirro EC. Reduction in handgrip strength and electromyographic activity in women with breast cancer. J Back Musculoskelet Rehabil. 2018;31(3):447-452. doi: 10.3233/BMR-170848. PMID 28946542
- [Background] Gomes PR, Freitas Junior IF, da Silva CB, Gomes IC, Rocha AP, Salgado AS, do Carmo EM. Short-term changes in handgrip strength, body composition, and lymphedema induced by breast cancer surgery. Rev Bras Ginecol Obstet. 2014 Jun;36(6):244-50. doi: 10.1590/s0100-720320140005004. PMID 25099463
- [Derived] Tugral A, Bakar Y, Akyol M. Predictors of Upper Extremity Function in Breast Cancer Survivors. Physiother Res Int. 2025 Jul;30(3):e70082. doi: 10.1002/pri.70082. PMID 40543072